CLINICAL TRIAL: NCT05777668
Title: A Predictive Nomogram for Trismus After Radiotherapy for Head and Neck Cancer
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4641
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Trismus
Keywords: radiation induced trismus, head and neck radiotherapy
MeSH Terms: conditions — Trismus | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Head and neck cancer patients undergoing radiotherapy
  Interventions: Radiation: Volumetric modulated radiotherapy

INTERVENTIONS:
Radiation: Volumetric modulated radiotherapy

SUMMARY:
Background: The aim of this study is to develop a prediction model for radiation-induced trismus (maximal interincisal distance equal to or less than 35 mm) based on a multivariable analysis of dosimetric and clinical factors.

DETAILED DESCRIPTION:
The maximum inter-incisal opening (MIO) of hean and neck cancer (HNC) patients who undergo radiotherapy (RT) ± concurrent chemotherapy with radical intent, will be prospectively measured prior to RT (baseline) and 6 months post-RT.

The potential risk factors (clinical and dosimetric) will be first screened by univariate analysis and then by multivariate analysis. At the end of this process, the features identified as relevant, will be used to fit a logistic regression model and calculate the probability of observed trismus during the 6-month follow-up after RT

ELIGIBILITY:
Inclusion Criteria:

* HNC
* treatment definitive or postoperative external beam radiotherapy, either alone or in -combination with chemotherapy or cetuximab at least 6 months follow-up

Exclusion Criteria:

* primary tumor out-side the head and neck region, intracranially, or if it originated from the nasal vestibule
* patient death during RT or within the first 6 months after the start of RT, no outcome data available

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with HNC treated consecutively with definitive or postoperative external beam radiotherapy, either alone or in combination with chemotherapy or cetuximab, between January 2017 and April 2021 at Gemelli Advanced Radiation Therapy (ART) center, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Trismus | 6 months
  maximal interincisal distance equal to or less than 35 mm

CONTACTS AND LOCATIONS:
Overall Officials: Mariangela Massaccesi, MD, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli

IPD SHARING:
Plan to Share IPD: Undecided